CLINICAL TRIAL: NCT02676089
Title: A 52 WEEK, RANDOMIZED, DOUBLE BLIND, MULTINATIONAL, MULTICENTRE, ACTIVE CONTROLLED, 3-ARM PARALLEL GROUP TRIAL COMPARING CHF 5993 200/6/12.5 µg pMDI (FIXED COMBINATION OF EXTRAFINE BECLOMETASONE DIPROPIONATE PLUS FORMOTEROL FUMARATE PLUS GLYCOPYRRONIUM BROMIDE) TO CHF 1535 200/6 µg pMDI (FIXED COMBINATION OF EXTRAFINE BECLOMETHASONE DIPROPIONATE PLUS FORMOTEROL FUMARATE) ALONE OR ON TOP OF OPEN-LABEL TIOTROPIUM 2.5 µg RESPIMAT® IN PATIENTS WITH ASTHMA UNCONTROLLED ON HIGH DOSES OF INHALED CORTICOSTEROIDS IN COMBINATION WITH LONG-ACTING ß2-AGONISTS
Brief Title: TRIple in Asthma hiGh strenGth vErsus Ics/Laba hs and tiotRopium (TRIGGER)
Acronym: TRIGGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-05993AB2-02; 2015-000717-40 (EudraCT Number)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Asthma, Anticholinergics, Triple combination
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CHF 5993 200/6/12.5 µg (Experimental): Treatment A:
  CHF 5993 200/6/12.5 µg: 2 inhalations bid Total daily dose: 800/24/50 µg BDP/FF/GB
  Interventions: Drug: CHF 5993 200/6/12.5 µg
- CHF 1535 200/6 µg (Active Comparator): Treatment B:
  CHF 1535 200/6 µg: 2 inhalations bid Total daily dose: 800/24 µg BDP/FF
  Interventions: Drug: CHF 1535 200/6 µg
- CHF 1535 200/6 µg + Tiotropium Respimat 2.5 µg (Active Comparator): Treatment C (open-label arm):
  CHF 1535 200/6 µg: 2 inhalations bid
  + Tiotropium Respimat 2.5 µg: 2 inhalations od Total daily dose: 800/24 µg BDP/FF + 5 µg Tio
  Interventions: Drug: CHF 1535 200/6 µg + Tiotropium Respimat 2.5 µg

INTERVENTIONS:
Drug: CHF 5993 200/6/12.5 µg
  Arms: CHF 5993 200/6/12.5 µg
Drug: CHF 1535 200/6 µg
  Arms: CHF 1535 200/6 µg
Drug: CHF 1535 200/6 µg + Tiotropium Respimat 2.5 µg
  Arms: CHF 1535 200/6 µg + Tiotropium Respimat 2.5 µg

SUMMARY:
The purpose of this study is to evaluate the superiority of CHF 5993 200/6/12.5 µg pMDI (fixed combination of extrafine beclometasone dipropionate plus formoterol fumarate plus glycopyrronium bromide) versus CHF 1535 200/6 µg pMDI (fixed combination of extrafine beclometasone dipropionate plus formoterol fumarate) and to compare the effect of CHF 5993 200/6/12.5 µg pMDI vs CHF 5993 200/6/12.5 µg plus open-label Tiotropium 2.5µg, in terms of lung functions parameters and rate of exacerbations, as well as to assess its safety and some health economics outcomes.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma ≥ 1 year and diagnosed before 40 years old
* Uncontrolled asthma with double therapy only on high doses of Inhaled CorticoSteroid (ICS) in combination with Long-Acting Beta2 Agonist (LABA) with ACQ-7 (Asthma Control Questionnaire) ≥1.5
* Pre-bronchodilator FEV1 <80% of the predicted normal value
* Positive reversibility test
* At least 1 documented asthma exacerbation in the previous year

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Patients with any asthma exacerbation or respiratory tract infection in the 4 weeks prior screening
* Current smoker or ex-smoker (>= 10 packs year)
* Any change in dose, schedule or formulation of ICS + LABA combination in the 4 weeks prior screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1433 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Pre-dose FEV1 (Forced Expiratory Volume in the first second) | Week 26
Reduction of moderate and severe asthma exacerbations rate | Week 0 to Week 52

SECONDARY OUTCOMES:
Peak FEV1 (Peak of Forced Expiratory Volume in the first second) within 3 hours post-dose | Week 26
Change from baseline in morning PEF (Peak Expiratory Flow) | Week 0 to Week 26
Reduction of severe asthma exacerbations rate | Week 0 to week 52
  Pooled analysis of CCD-05993AB1-03 and CCD-05993AB2-02 trials

OTHER OUTCOMES:
Adverse Events and Adverse Drug reactions | Up to Week 52
Collection of Health Economics outcomes | Week 0 to Week 52
  Total use of healthcare resources and absence from work

CONTACTS AND LOCATIONS:
Overall Officials: Georgio Walter Canonica, MD, Principal Investigator — University of Medicine, Genoa, Italy
Locations (244):
- Argentina (6):
  - Chiesi Clinical Trial Site 432702, Buenos Aires
  - Chiesi Clinical Trial Site 432704, CABA
  - Chiesi Clinical Trial Site 432705, Mar del Plata
  - Chiesi Clinical Trial Site 432701, Quilmes
  - Chiesi Clinical Trial Site 432703, San Miguel de Tucumán
  - Chiesi Clinical Trial Site 432706, San Miguel de Tucumán
- Belarus (5):
  - Chiesi Clinical Trial Site 112703, Homyel
  - Chiesi Clinical Trial Site 112704, Homyel
  - Chiesi Clinical Trial Site 112701, Minsk
  - Chiesi Clinical Trial Site 112702, Minsk
  - Chiesi Clinical Trial Site 112705, Minsk
- Bulgaria (20):
  - Chiesi Clinical Trial Site 100707, Blagoevgrad
  - Chiesi Clinical Trial Site 100720, Burgas
  - Chiesi Clinical Trial Site 100718, Gabrovo
  - Chiesi Clinical Trial Site 100713, Haskovo
  - Chiesi Clinical Trial Site 100722, Montana
  - Chiesi Clinical Trial Site 100702, Pleven
  - Chiesi Clinical Trial Site 100705, Plovdiv
  - Chiesi Clinical Trial Site 100708, Plovdiv
  - Chiesi Clinical Trial Site 100715, Plovdiv
  - Chiesi Clinical Trial Site 100716, Rousse
  - Chiesi Clinical Trial Site 100701, Sofia
  - Chiesi Clinical Trial Site 100703, Sofia
  - Chiesi Clinical Trial Site 100704, Sofia
  - Chiesi Clinical Trial Site 100709, Sofia
  - Chiesi Clinical Trial Site 100719, Sofia
  - Chiesi Clinical Trial Site 100706, Stara Zagora
  - Chiesi Clinical Trial Site 100712, Stara Zagora
  - Chiesi Clinical Trial Site 100710, Varna
  - Chiesi Clinical Trial Site 100711, Vidin
  - Chiesi Clinical Trial Site 100721, Vidin
- Czechia (13):
  - Chiesi Clinical Trial Site 203711, Blansko
  - Chiesi Clinical Trial Site 203702, Brandýs nad Labem
  - Chiesi Clinical Trial Site 203708, Brno
  - Chiesi Clinical Trial Site 203707, Jindřichův Hradec
  - Chiesi Clinical Trial Site 203705, Kralupy nad Vltavou
  - Chiesi Clinical Trial Site 203709, Moravský Krumlov
  - Chiesi Clinical Trial Site 203704, Opava
  - Chiesi Clinical Trial Site 203701, Prague
  - Chiesi Clinical Trial Site 203703, Prague
  - Chiesi Clinical Trial Site 203710, Prague
  - Chiesi Clinical Trial Site 203713, Rokycany
  - Chiesi Clinical Trial Site 203706, Teplice
  - Chiesi Clinical Trial Site 203712, Varnsdorf
- Germany (15):
  - Chiesi Clinical Trial Site 276709, Berlin
  - Chiesi Clinical Trial Site 276712, Berlin
  - Chiesi Clinical Trial Site 276711, Bonn
  - Chiesi Clinical Trial Site 276707, Frankfurt am Main
  - Chiesi Clinical Trial Site 276714, Frankfurt am Main
  - Chiesi Clinical Trial Site 276705, Hamburg
  - Chiesi Clinical Trial Site 276703, Hanover
  - Chiesi Clinical Trial Site 276708, Koblenz
  - Chiesi Clinical Trial Site 276702, Leipzig
  - Chiesi Clinical Trial Site 276704, Leipzig
  - Chiesi Clinical Trial Site 276710, Leipzig
  - Chiesi Clinical Trial Site 276715, Mainz
  - Chiesi Clinical Trial Site 276701, München
  - Chiesi Clinical Trial Site 276713, Münster
  - Chiesi Clinical Trial Site 276716, Rosenheim
- Hungary (19):
  - Chiesi Clinical Trial Site 348707, Balassagyarmat
  - Chiesi Clinical Trial Site 348715, Budapest
  - Chiesi Clinical Trial Site 348721, Debrecen
  - Chiesi Clinical Trial Site 348708, Érd
  - Chiesi Clinical Trial Site 348712, Gödöllő
  - Chiesi Clinical Trial Site 348718, Hatvan
  - Chiesi Clinical Trial Site 348717, Komárom
  - Chiesi Clinical Trial Site 348709, Létavértes
  - Chiesi Clinical Trial Site 348703, Monor
  - Chiesi Clinical Trial Site 348719, Mórahalom
  - Chiesi Clinical Trial Site 348704, Nyíregyháza
  - Chiesi Clinical Trial Site 348714, Nyíregyháza
  - Chiesi Clinical Trial Site 348713, Pécs
  - Chiesi Clinical Trial Site 348702, Siófok
  - Chiesi Clinical Trial Site 348706, Szarvas
  - Chiesi Clinical Trial Site 348701, Szeged
  - Chiesi Clinical Trial Site 348705, Szentgotthárd
  - Chiesi Clinical Trial Site 348710, Vásárosnamény
  - Chiesi Clinical Trial Site 348720, Vecsés
- Italy (6):
  - Chiesi Clinical Trial Site 380704, Bologna
  - Chiesi Clinical Trial Site 380703, Catania
  - Chiesi Clinical Trial Site 380701, Genova
  - Chiesi Clinical Trial Site 380705, Palermo
  - Chiesi Clinical Trial Site 380702, Pavia
  - Chiesi Clinical Trial Site 380706, Tradate
- Lithuania (4):
  - Chiesi Clinical Trial Site 440701, Šiauliai
  - Chiesi Clinical Trial Site 440702, Vilnius
  - Chiesi Clinical Trial Site 440703, Vilnius
  - Chiesi Clinical Trial Site 440705, Vilnius
- Poland (34):
  - Chiesi Clinical Trial Site 616713, Bialystok
  - Chiesi Clinical Trial Site 616718, Bialystok
  - Chiesi Clinical Trial Site 616722, Bielsko-Biala
  - Chiesi Clinical Trial Site 616702, Bienkówka
  - Chiesi Clinical Trial Site 616727, Bydgoszcz
  - Chiesi Clinical Trial Site 616701, Gdansk
  - Chiesi Clinical Trial Site 616704, Giżycko
  - Chiesi Clinical Trial Site 616716, Grudziądz
  - Chiesi Clinical Trial Site 616725, Katowice
  - Chiesi Clinical Trial Site 616729, Katowice
  - Chiesi Clinical Trial Site 616719, Krakow
  - Chiesi Clinical Trial Site 616734, Krakow
  - Chiesi Clinical Trial Site 616736, Krakow
  - Chiesi Clinical Trial Site 616707, Lodz
  - Chiesi Clinical Trial Site 616708, Lodz
  - Chiesi Clinical Trial Site 616711, Lodz
  - Chiesi Clinical Trial Site 616726, Lodz
  - Chiesi Clinical Trial Site 616733, Mrozy
  - Chiesi Clinical Trial Site 616717, Ostróda
  - Chiesi Clinical Trial Site 616731, Otwock
  - Chiesi Clinical Trial Site 616703, Pabianice
  - Chiesi Clinical Trial Site 616709, Poznan
  - Chiesi Clinical Trial Site 616728, Poznan
  - Chiesi Clinical Trial Site 616720, Proszowice
  - Chiesi Clinical Trial Site 616723, Rzeszów
  - Chiesi Clinical Trial Site 616735, Rzeszów
  - Chiesi Clinical Trial Site 616721, Skierniewice
  - Chiesi Clinical Trial Site 616732, Strzelce Opolskie
  - Chiesi Clinical Trial Site 616712, Świdnik
  - Chiesi Clinical Trial Site 616710, Tarnów
  - Chiesi Clinical Trial Site 616730, Wilkowice
  - Chiesi Clinical Trial Site 616705, Wroclaw
  - Chiesi Clinical Trial Site 616714, Wroclaw
  - Chiesi Clinical Trial Site 616715, Wroclaw
- Portugal (5):
  - Chiesi Clinical Trial Site 620704, Aveiro
  - Chiesi Clinical Trial Site 620703, Figueira da Foz Municipality
  - Chiesi Clinical Trial Site 620702, Lisbon
  - Chiesi Clinical Trial Site 620708, Loures
  - Chiesi Clinical Trial Site 620707, Vila Nova de Gaia
- Romania (21):
  - Chiesi Clinical Trial Site 642715, Alexandru cel Bun
  - Chiesi Clinical Trial Site 642713, Arad
  - Chiesi Clinical Trial Site 642722, Bacau
  - Chiesi Clinical Trial Site 642717, Bragadiru
  - Chiesi Clinical Trial Site 642706, Brasov
  - Chiesi Clinical Trial Site 642703, Bucharest
  - Chiesi Clinical Trial Site 642707, Bucharest
  - Chiesi Clinical Trial Site 642708, Bucharest
  - Chiesi Clinical Trial Site 642719, Bucharest
  - Chiesi Clinical Trial Site 642723, Bucharest
  - Chiesi Clinical Trial Site 642709, Cluj-Napoca
  - Chiesi Clinical Trial Site 642714, Cluj-Napoca
  - Chiesi Clinical Trial Site 642716, Cluj-Napoca
  - Chiesi Clinical Trial Site 642718, Cluj-Napoca
  - Chiesi Clinical Trial Site 642726, Cluj-Napoca
  - Chiesi Clinical Trial Site 642712, Craiova
  - Chiesi Clinical Trial Site 642704, Iași
  - Chiesi Clinical Trial Site 642710, Iași
  - Chiesi Clinical Trial Site 642705, Oradea
  - Chiesi Clinical Trial Site 642711, Suceava
  - Chiesi Clinical Trial Site 642721, Timișoara
- Russia (53):
  - Chiesi Clinical Trial Site 643724, Anton
  - Chiesi Clinical Trial Site 643727, Chelyabinsk
  - Chiesi Clinical Trial Site 643733, Chelyabinsk
  - Chiesi Clinical Trial Site 643745, Chelyabinsk
  - Chiesi Clinical Trial Site 643754, Izhevsk
  - Chiesi Clinical Trial Site 643713, Kazan'
  - Chiesi Clinical Trial Site 643719, Kazan'
  - Chiesi Clinical Trial Site 643741, Kazan'
  - Chiesi Clinical Trial Site 643746, Kazan'
  - Chiesi Clinical Trial Site 643704, Kemerovo
  - Chiesi Clinical Trial Site 643731, Kemerovo
  - Chiesi Clinical Trial Site 643702, Moscow
  - Chiesi Clinical Trial Site 643705, Moscow
  - Chiesi Clinical Trial Site 643706, Moscow
  - Chiesi Clinical Trial Site 643718, Moscow
  - Chiesi Clinical Trial Site 643722, Moscow
  - Chiesi Clinical Trial Site 643735, Moscow
  - Chiesi Clinical Trial Site 643743, Moscow
  - Chiesi Clinical Trial Site 643707, Nizhny Novgorod
  - Chiesi Clinical Trial Site 643723, Nizhny Novgorod
  - Chiesi Clinical Trial Site 643744, Nizhny Novgorod
  - Chiesi Clinical Trial Site 643717, Novosibirsk
  - Chiesi Clinical Trial Site 643729, Orenburg
  - Chiesi Clinical Trial Site 643711, Pyatigorsk
  - Chiesi Clinical Trial Site 643701, Ryazan
  - Chiesi Clinical Trial Site 643712, Saint Petersburg
  - Chiesi Clinical Trial Site 643714, Saint Petersburg
  - Chiesi Clinical Trial Site 643715, Saint Petersburg
  - Chiesi Clinical Trial Site 643716, Saint Petersburg
  - Chiesi Clinical Trial Site 643725, Saint Petersburg
  - Chiesi Clinical Trial Site 643730, Saint Petersburg
  - Chiesi Clinical Trial Site 643732, Saint Petersburg
  - Chiesi Clinical Trial Site 643737, Saint Petersburg
  - Chiesi Clinical Trial Site 643739, Saint Petersburg
  - Chiesi Clinical Trial Site 643752, Saint Petersburg
  - Chiesi Clinical Trial Site 643757, Saint Petersburg
  - Chiesi Clinical Trial Site 643758, Saint Petersburg
  - Chiesi Clinical Trial Site 643703, Saratov
  - Chiesi Clinical Trial Site 643736, Saratov
  - Chiesi Clinical Trial Site 643726, Smolensk
  - Chiesi Clinical Trial Site 643740, Stavropol
  - Chiesi Clinical Trial Site 643709, Tomsk
  - Chiesi Clinical Trial Site 643728, Tomsk
  - Chiesi Clinical Trial Site 643759, Tomsk
  - Chiesi Clinical Trial Site 643755, Ufa
  - Chiesi Clinical Trial Site 643708, Vladikavkaz
  - Chiesi Clinical Trial Site 643738, Vladimir
  - Chiesi Clinical Trial Site 643710, Voronezh
  - Chiesi Clinical Trial Site 643720, Yaroslavl
  - Chiesi Clinical Trial Site 643734, Yaroslavl
  - Chiesi Clinical Trial Site 643742, Yaroslavl
  - Chiesi Clinical Trial Site 643749, Yaroslavl
  - Chiesi Clinical Trial Site 643721, Yekaterinburg
- Slovakia (9):
  - Chiesi Clinical Trial Site 703704, Bratislava
  - Chiesi Clinical Trial Site 703707, Bratislava
  - Chiesi Clinical Trial Site 703702, Ilava
  - Chiesi Clinical Trial Site 703705, Košice
  - Chiesi Clinical Trial Site 703706, Košice
  - Chiesi Clinical Trial Site 703701, Nové Zámky
  - Chiesi Clinical Trial Site 703709, Prievidza
  - Chiesi Clinical Trial Site 703703, Spišská Nová Ves
  - Chiesi Clinical Trial Site 703708, Štúrovo
- Spain (7):
  - Chiesi Clinical Trial Site 724702, A Coruña
  - Chiesi Clinical Trial Site 724703, Badajoz
  - Chiesi Clinical Trial Site 724706, Badalona
  - Chiesi Clinical Trial Site 724701, Madrid
  - Chiesi Clinical Trial Site 724704, Madrid
  - Chiesi Clinical Trial Site 724705, Málaga
  - Chiesi Clinical Trial Site 724707, Sabadell
- Turkey (Türkiye) (9):
  - Chiesi Clinical Trial Site 792701, Ankara
  - Chiesi Clinical Trial Site 792702, Ankara
  - Chiesi Clinical Trial Site 792703, Antalya
  - Chiesi Clinical Trial Site 792710, Aydin
  - Chiesi Clinical Trial Site 792707, Istanbul
  - Chiesi Clinical Trial Site 792706, Kocaeli
  - Chiesi Clinical Trial Site 792705, Maltepe
  - Chiesi Clinical Trial Site 792708, Mersin
  - Chiesi Clinical Trial Site 792709, Yenişehir
- Ukraine (14):
  - Chiesi Clinical Trial Site 804701, Dnipro
  - Chiesi Clinical Trial Site 804711, Ivano-Frankivsk
  - Chiesi Clinical Trial Site 804709, Kharkiv
  - Chiesi Clinical Trial Site 804710, Kherson
  - Chiesi Clinical Trial Site 804713, Kiev
  - Chiesi Clinical Trial Site 804705, Kyiv
  - Chiesi Clinical Trial Site 804712, Lviv
  - Chiesi Clinical Trial Site 804715, Sumy
  - Chiesi Clinical Trial Site 804703, Vinnytsia
  - Chiesi Clinical Trial Site 804706, Vinnytsia
  - Chiesi Clinical Trial Site 804707, Vinnytsia
  - Chiesi Clinical Trial Site 804714, Vinnytsia
  - Chiesi Clinical Trial Site 804704, Zaporizhzhya
  - Chiesi Clinical Trial Site 804708, Zhytomyr
- United Kingdom (4):
  - Chiesi Clinical Trial Site 826702, Llanelli
  - Chiesi Clinical Trial Site 826703, London
  - Chiesi Clinical Trial Site 826704, Manchester
  - Chiesi Clinical Trial Site 826701, Soham

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Result] Virchow JC, Kuna P, Paggiaro P, Papi A, Singh D, Corre S, Zuccaro F, Vele A, Kots M, Georges G, Petruzzelli S, Canonica GW. Single inhaler extrafine triple therapy in uncontrolled asthma (TRIMARAN and TRIGGER): two double-blind, parallel-group, randomised, controlled phase 3 trials. Lancet. 2019 Nov 9;394(10210):1737-1749. doi: 10.1016/S0140-6736(19)32215-9. Epub 2019 Sep 30. PMID 31582314
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Orlovic M, Magni T, Lukyanov V, Guerra I, Madoni A. Cost-effectiveness of single-inhaler extrafine beclometasone dipropionate/formoterol fumarate/glycopyrronium in patients with uncontrolled asthma in England. Respir Med. 2022 Sep;201:106934. doi: 10.1016/j.rmed.2022.106934. Epub 2022 Jul 19. PMID 35872377
- [Derived] Papi A, Singh D, Virchow JC, Canonica GW, Vele A, Georges G. Normalisation of airflow limitation in asthma: Post-hoc analyses of TRIMARAN and TRIGGER. Clin Transl Allergy. 2022 Apr 17;12(4):e12145. doi: 10.1002/clt2.12145. eCollection 2022 Apr. PMID 35450196
- [Derived] Singh D, Virchow JC, Canonica GW, Vele A, Kots M, Georges G, Papi A. Determinants of response to inhaled extrafine triple therapy in asthma: analyses of TRIMARAN and TRIGGER. Respir Res. 2020 Oct 29;21(1):285. doi: 10.1186/s12931-020-01558-y. PMID 33121501
- [Derived] Singh D, Virchow JC, Canonica GW, Vele A, Kots M, Georges G, Papi A. Extrafine triple therapy in patients with asthma and persistent airflow limitation. Eur Respir J. 2020 Sep 24;56(3):2000476. doi: 10.1183/13993003.00476-2020. Print 2020 Sep. No abstract available. PMID 32430414
- See also: Study Record on EU Clinical Trials Register including results. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-000717-40/results